CLINICAL TRIAL: NCT01358019
Title: A Phase 1 Study of LY2523355 in Patients With Solid Cancer
Brief Title: A Study of LY2523355 in Patients With Solid Cancer
Acronym: 2523355-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2523355-001
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — litronesib

ARMS (1):
- LY2523355 (Experimental)
  Interventions: Drug: LY2523355

INTERVENTIONS:
Drug: LY2523355 — Days 1, 2, and 3 in a cycle that consists of 21-days

SUMMARY:
The primary objective of this study is to examine a recommended dose for subsequent phase trial(s), by the observation of the safety and toxicity profiles of LY2523355 in patients with advanced and/or metastatic cancer. The secondary objectives are to study the pharmacokinetics and antitumor effect.

ELIGIBILITY:
Inclusion Criteria:

* Histological and/or cytological evidence of solid tumors
* A diagnosis of advanced and/or metastatic solid tumors
* Patients who are refractory to standard therapy or for which no proven effective therapy exists
* Written informed consent
* Appropriate bone marrow, hepatic and renal functions
* ECOG PS =< 1

Exclusion Criteria:

* Have serious preexisting complication
* Have active infection which requires intravenous antibiotics
* Have symptomatic central nervous system metastases
* Have current acute or chronic leukemia
* Have had an autologous or allogenic hematopoietic stem cell transplantation
* Have active multiple cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity based on the Common Terminology Criteria for Adverse Events v4.0
Number of patients with adverse events

SECONDARY OUTCOMES:
Pharmacokinetics
  Plasma concentration of LY2523355 and metabolite
Antitumor effect
  Response evaluation criteria in solid tumors

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Wakui H, Yamamoto N, Kitazono S, Mizugaki H, Nakamichi S, Fujiwara Y, Nokihara H, Yamada Y, Suzuki K, Kanda H, Akinaga S, Tamura T. A phase 1 and dose-finding study of LY2523355 (litronesib), an Eg5 inhibitor, in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2014 Jul;74(1):15-23. doi: 10.1007/s00280-014-2467-z. Epub 2014 Apr 22. PMID 24752449